CLINICAL TRIAL: NCT04359017
Title: Systemic Absorption of Lidocaine After Ultrasound Guided Hematoma Block for Reduction of Different Types of Pediatric Distal Radius Fractures
Brief Title: Systemic Absorption of Lidocaine After Hematoma Block
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsoring staff have left institution
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202004180
Record Dates: First submitted 2020-04-17; First posted 2020-04-24 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Radius Fracture Distal; Hematoma; Lidocaine; Pediatrics
MeSH Terms: conditions — Wrist Fractures; Hematoma | interventions — Lidocaine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lidocaine Hematoma Block (Experimental)
  Interventions: Drug: Lidocaine 1% Injectable Solution

INTERVENTIONS:
Drug: Lidocaine 1% Injectable Solution — The lidocaine will be injected into the fracture hematoma using buffered 1% lidocaine solution at a dose of 2.5 mg/kg (0.25 mL/kg), maximum dose 100 mg (10 mL). Using a 30-gauge needle to minimize pain, a small skin wheal of lidocaine will be injected over the fracture site. A 21-gauge needle will then be attached to the lidocaine filled syringe and passed through the skin wheal used to inject the lidocaine into the fracture hematoma. To confirm the needle is in the fracture hematoma, a small amount of blood from the hematoma will be aspirated into the syringe filled with lidocaine before injecting the lidocaine, as in standard practice.

SUMMARY:
This study will measure in children how much numbing medicine, lidocaine, is absorbed into the bloodstream after it is injected into a blood clot (hematoma) around a forearm fracture for pain control when the broken bone is moved back into place (fracture reduction). This is called a hematoma block and is commonly used in the Emergency Unit. To help with anxiety and to add additional pain control, nitrous oxide (laughing gas) is given while the lidocaine hematoma block is placed and continued during the fracture reduction. Advantages of using this technique for pain control instead of an intravenous anesthetic such as ketamine include faster recovery and discharge home, and longer pain control.

Of concern, if too much lidocaine is absorbed into the bloodstream, seizures and irregular heart beating may occur. Bloodstream concentrations of lidocaine after a hematoma block have been measured in only one study of 8 adults and found to be at significant but safe levels. No study has been published in children to measure bloodstream lidocaine levels when a hematoma block is used. Because children's bones are still growing and more metabolically active than adult bones, the investigators believe it is important to determine whether lidocaine blood levels in children are also at safe levels when using a standard lidocaine hematoma block for reduction of fractures. The investigators also want to determine whether bloodstream lidocaine levels correlate with type of fracture.

The investigators also aim to determine if there is a difference in absorption pattern between different types of distal radius fractures, if there is a correlation between fracture type and systemic lidocaine absorption, and if there is a correlation between fracture type and ability to provide adequate pain and sedation control with lidocaine hematoma block/inhaled nitrous combination. The investigators believe blood lidocaine levels after hematoma block in children will peak at safe levels, but will be higher than those observed in adults.

DETAILED DESCRIPTION:
When a subject with an eligible distal forearm fracture is identified, the subject will be approached for enrollment and consent.

50% nitrous oxide/50% oxygen then will be administered to the subject by face mask for a minimum of 2 minutes before venous catheter insertion (50% nitrous oxide will continue to be administered until fracture reduction is completed). Nitrous oxide currently is administered regularly in the St. Louis Children's Emergency Department for painful procedures including fracture reduction, abscess incision and drainage, laceration repair and venous catheter placement. Nitrous oxide 50% blended with 50% oxygen will be administered for this study by credentialed emergency unit staff using a continuous flow delivery system that includes scavenging of exhaled nitrous oxide. Standard monitoring for deep sedation will be used as described in the clinical protocol.

A venous catheter then will be inserted into the uninjured arm. A lidocaine hematoma block will be injected under ultrasound guidance by a pediatric emergency medicine physician using 2.5 mg/kg, maximum of 100mg, of 1% buffered lidocaine. The recommended lidocaine dose for hematoma block in children is 3-5 mg/kg. However, in a previous study, in another pediatric trial, and in the single report of plasma lidocaine levels in adults, 2.5 mg/kg of 1% lidocaine based upon the patient's weight, maximum 100 mg, was found effective and without adverse effects. The Pediatric Sedation State Scale will be administered by the sedation provider, and a research assistant when available, and used to determine if pain control is adequate, or if rescue IV analgesia is needed. This scale has been validated for procedural sedation.

Serial blood samples will be drawn through the indwelling venous catheter by a nurse or medic at 5, 10, 20, 40 and 60 minutes after injection of the hematoma block. Serial plasma lidocaine levels will be measured as follows. 5 mL samples of blood will be obtained via the indwelling venous catheter at 5, 10, 20, 40 and 60 minutes after injection of the lidocaine hematoma block. The samples of blood will be collected in standard red top vacutainer blood tubes and processed, frozen and stored in the SLCH/BJC Lab.

At 5 minutes after the hematoma block injection, the orthopedic surgeon will attempt fracture reduction. If the subject has minimal response to squeezing the fracture site prior to 5 minutes post injection, reduction may begin at that time. Nitrous oxide administration will be stopped and administration of 100% oxygen will begin when the orthopedic surgeon indicates satisfactory fracture reduction as determined by bedside fluoroscopy (standard procedure), a cast or splint has been applied, and, if necessary, the cast has been split. Oxygen administration will be stopped when the subject's exhaled nitrous oxide concentration falls below 10% or the subject pulls the nitrous oxide mask off the face.

If the subject resists the fracture reduction, verbally indicates significant pain, or has an unfavorable PSSS, ketamine sedation will be administered via the indwelling venous catheter and fracture reduction completed under deep sedation. Post procedure pain score via the Wong-Baker Faces scale, and post procedure surveys will be administered 15 minutes after nitrous administration is stopped. After the subject's recovery from sedation, the subject, subject's parents/guardians, physician providing sedation (inhaled nitrous) and the orthopedic surgeon will be asked to rate their satisfaction with the sedation and analgesia for the fracture reduction using a Likert scale ranging from 1 (not satisfied at all) to 10 (very satisfied). Recovery from sedation satisfactory for discharge home is indicated by a score of 10 on the Modified Aldrete Scale below, and the child can sit up unaided along with control of pain and vomiting. Family will be contacted via telephone 48 hours after their visit to assess for any late adverse effects.

Adverse events will be documented on a data collection sheet using consensus-based definitions that include the event, time and any intervention employed. In addition, the subject will be asked about symptoms typically seen with procedural sedation and lidocaine toxicity including: vomiting, nausea, tinnitus, circumoral or tongue numbness, metallic taste in mouth, nystagmus, vision changes, muscle twitching, tremors, seizure, respiratory depression, chest pain, difficulty breathing, palpitations, ECG changes on monitor (type noted, ECG strip printed), and any other unpleasant or euphoric symptom.

ELIGIBILITY:
Inclusion Criteria:

* ASA status class 1 or 2
* Ages 5-17
* Parent/guardian is present

Exclusion Criteria:

* Open fracture
* Previous attempt at reduction
* Multiple other injuries
* Physeal (growth plate) fractures
* Volar displacement of the distal fracture fragment
* Delayed presentation (>48 hrs from injury)
* Concern for significant neurovascular injury
* Refracture through a healing fracture
* History of adverse effect from lidocaine or nitrous oxide
* Active psychosis
* Non English speaking parents
* Liver disease
* Cardiac disease
* Abnormal bones such as osteogenesis imperfecta or osteopenia from lack of use
* Developmental abnormalities

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Plasma Lidocaine Levels | Serial plasma lidocaine levels will be measured during a single subject's distal forearm fracture reduction, to be measured over the course of 60 minutes form the injection of lidocaine into the hematoma block.
  Measured concentrations of plasma lidocaine levels for subjects undergoing lidocaine hematoma block for their distal radius fracture reduction.

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Louis Children's Hospital, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bear DM, Friel NA, Lupo CL, Pitetti R, Ward WT. Hematoma block versus sedation for the reduction of distal radius fractures in children. J Hand Surg Am. 2015 Jan;40(1):57-61. doi: 10.1016/j.jhsa.2014.08.039. Epub 2014 Oct 11. PMID 25306504
- [Background] Blasier RD. Anesthetic considerations for fracture management in the outpatient setting. J Pediatr Orthop. 2004 Nov-Dec;24(6):742-6. doi: 10.1097/00004694-200411000-00027. No abstract available. PMID 15502581
- [Background] Cote CJ, Wilson S. Guidelines for Monitoring and Management of Pediatric Patients Before, During, and After Sedation for Diagnostic and Therapeutic Procedures. Pediatr Dent. 2019 Jul 15;41(4):26E-52E. PMID 31439094
- [Background] Cravero JP, Askins N, Sriswasdi P, Tsze DS, Zurakowski D, Sinnott S. Validation of the Pediatric Sedation State Scale. Pediatrics. 2017 May;139(5):e20162897. doi: 10.1542/peds.2016-2897. PMID 28557732
- [Background] Kennedy RM, Porter FL, Miller JP, Jaffe DM. Comparison of fentanyl/midazolam with ketamine/midazolam for pediatric orthopedic emergencies. Pediatrics. 1998 Oct;102(4 Pt 1):956-63. doi: 10.1542/peds.102.4.956. PMID 9755272
- [Background] Luhmann JD, Schootman M, Luhmann SJ, Kennedy RM. A randomized comparison of nitrous oxide plus hematoma block versus ketamine plus midazolam for emergency department forearm fracture reduction in children. Pediatrics. 2006 Oct;118(4):e1078-86. doi: 10.1542/peds.2005-1694. Epub 2006 Sep 11. PMID 16966390
- [Background] Meinig RP, Quick A, Lobmeyer L. Plasma lidocaine levels following hematoma block for distal radius fractures. J Orthop Trauma. 1989;3(3):187-91. doi: 10.1097/00005131-198909000-00001. PMID 2809817
- [Background] Naranje SM, Erali RA, Warner WC Jr, Sawyer JR, Kelly DM. Epidemiology of Pediatric Fractures Presenting to Emergency Departments in the United States. J Pediatr Orthop. 2016 Jun;36(4):e45-8. doi: 10.1097/BPO.0000000000000595. PMID 26177059